CLINICAL TRIAL: NCT04154176
Title: Validation of the Greek Version of the Confusion Assessment Method Diagnostic Algorithm (CAM) and the Nursing Delirium Screening Scale (Nu-DESC) and Their Inter-rater Reliablity: A Prospective Cohort Study
Brief Title: Validation of the Greek Version of the Confusion Assessment Method Diagnostic Algorithm (CAM) and the Nursing Delirium Screening Scale (Nu-DESC) and Their Inter-rater Reliablity
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: CAM Nu-DESC in Greek
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POD CAM Nu-DESC: Patients undergoing surgery under general anesthesia assessed for POD with CAM and Nu-DESC
  Interventions: Other: CAM, Nu-DESC

INTERVENTIONS:
Other: CAM, Nu-DESC — Two trained raters, who are blinded and have no access to each other's evaluation, administer the CAM and Nu-DESC questionnaires in each shift, during the first postoperative day after the discharge from the post-anaesthesia care unit, independently. The two assessments are completed within 60 minutes of each other. If the research team set the diagnosis of POD, the appropriate treatment will be initiated, according to the Hospital's protocol

SUMMARY:
This study attempts to validate the Greek version of the CAM Diagnostic Algorithm and Nu-DESC in patients undergoing surgery under general anesthesia.

DETAILED DESCRIPTION:
Accurate diagnosis for Greek speaking patients suffering from postoperative delirium is limited by the need for a translation of standardized tools that were investigated for their inter-rater reliability/agreement.

Our primary aim is to validate the Greek version of the CAM Diagnostic Algorithm and Nu-DESC in patients undergoing surgery under general anesthesia. Our secondary aim is to estimate the diagnostic accuracy of NuDESK in our population.

This study will provide the first official Greek translation of CAM and Nu-DESC, according to the ISPOR guidelines, and the first evaluation of their inter-rater agreement.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients over 60 years of age
2. an American Society of Anesthesiologists (ASA) physical status I to III
3. undergoing elective non-cardiac surgery under general anaesthesia
4. native speakers of the Greek language
5. eligible to leave the post-anaesthesia care unit
6. an expected in-hospital stay of at least 24 hours following surgery

Exclusion Criteria:

1. refused to participate or sign the informed consent form
2. surgery or anaesthesia within the last 30 day
3. any prior or current history involving an affliction of the central nervous system
4. severe hearing or visual impairment
5. psychiatric disorders
6. sa core less than 5 according the Geriatric Depression Scale (GDS-15)
7. a score less than 4 for females and less than 2 for males according to the Lawton-Brody Instrumental Activities of Daily Living Scale (I.A.D.L.)
8. alcohol consumption less than 35 units/week
9. drug dependence
10. previous neuropsychological testing
11. haemodynamical instability
12. peri-procedural desaturation (one or more events of SpO2<80% for more than 2 minutes)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Validation of the Greek version of the CAM Diagnostic Algorithm and Nu-DESC | 1st postoperative day
  validate the Greek version of the CAM Diagnostic Algorithm and Nu-DESC

SECONDARY OUTCOMES:
Estimation of the inter-rater agreement of the Greek versions of the CAM and Nu-DESC | 1st postoperative day
  estimate the inter-rater agreement of the Greek versions of the CAM and Nu-DESC
Incidence of POD in our study sample. | 1st postoperative day
  Estimate the incidence of POD in our study sample.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly
Locations (1):
- Univeristy of Thessaly, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ntalouka MP, Bareka M, Brotis AG, Chalkias A, Stamoulis K, Flossos A, Tzimas P, Arnaoutoglou E. Translation and cultural adaptation of the Greek version of the confusion assessment method diagnostic algorithm and the nursing delirium screening scale and their inter-rater reliability: A prospective cohort study. Hippokratia. 2020 Jan-Mar;24(1):8-14. PMID 33364733